CLINICAL TRIAL: NCT05101642
Title: Guided Creeping Technique (GCT) as a Novel Minimally Invasive Approach in Treating Gingival Recession - Single Arm Preliminary Study
Brief Title: Guided Creeping Technique (GCT) in Treating Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, Professor of Periodontology, October 6 University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-21
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Gingival Recession
Keywords: Minimally Invasive Surgery; Tunneling Techniques; Gingival Recession; Creeping Attachment
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided Creeping Technique (GCT) (Experimental): Novel minimally invasive guided creeping technique
  Interventions: Procedure: Guided Creeping Technique (GCT)

INTERVENTIONS:
Procedure: Guided Creeping Technique (GCT) — Guided Creeping Technique (GCT) is a novel minimally invasive blind tunnel

SUMMARY:
A novel minimally invasive guided creeping technique (GCT) is suggested to treat gingival recessions.

DETAILED DESCRIPTION:
Background: Coronally advanced flap with connective tissue grafting in a conventional or minimally invasive approaches includes massive soft tissue reflection that reduce soft tissue support and compromise vascularity around the grafted material. In an attempt to preserve soft tissue support, graft stability and maximizing graft protection in treating recession defects the present novel minimally invasive guided creeping technique (GCT) is suggested.

Methods: Twelve patients, each contributing a single Cairo RT1 GR defect, were treated by guided creeping technique and completed the 6 months follow up. Clinical, evaluations were performed and differences among groups were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Systemically and periodontally healthy
* Presence of isolated buccal Cairo RT1 gingival recessions
* An identifiable CEJ
* Affected teeth with at least 2mm attached gingiva.

Exclusion Criteria:

* Smokers
* Pregnancy
* Using antiepileptic drugs
* Using antibiotics for at least 20 days before surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Recession Coverage | Change from baseline to 6 months
  Measured in mm

SECONDARY OUTCOMES:
Keratinized Tissue Width | Change from baseline to 6 months
  Measured in mm
Keratinized Tissue Thickness | Change from baseline to 6 months
  Measured in mm

OTHER OUTCOMES:
Patient Reported Outcome | Through 14 days
  Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, Professor, Principal Investigator — Faculty of Dentistry, October 6 University
Locations (1):
- October 6 University, Giza, Egypt